CLINICAL TRIAL: NCT04699253
Title: Usability and Feasibility of a Personalized, Web-based Education and Self-management Approach for Patients With Chronic Heart Failure Across Four European Sites
Acronym: STABILISE-HF
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: RWTH Aachen University (Other); Queen's University, Belfast (Other); University College Dublin (Other)
Responsible Party: Sponsor
Other Study IDs: NL75892.068.20; NWE702 (Other Grant/Funding Number: Interreg NWE)
Record Dates: First submitted 2020-12-16; First posted 2021-01-07 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; patient self-management; patient education; web application

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Consenting participants: Patients meeting the eligibility criteria and are using the SanaCoach heart failure during the study period.
  Interventions: Device: SanaCoach Heart failure
- Consenting non-participants: Patients meeting the eligibility criteria but do not wish to use the SanaCoach heart failure and only fill-in an anonymized questionnaire once, without any follow-up.

INTERVENTIONS:
Device: SanaCoach Heart failure — Patients will be using the SanaCoach heart failure for at least 6 months during the study period. SanaCoach heart failure is a web application that will be guiding the patient through a regular, systematic assessment of patient's health and wellbeing as well as regular education sessions. The assessment frequency ranges from daily to monthly, based on the settings provided by the health care provider. Furthermore, it provides a repository for patient's care plan to give insight into the course and treatment of the disorder and offers the possibility to contact the health care provider through the web application.
  Groups: Consenting participants

SUMMARY:
The STABELISE-HF is an investigator initiated, international, multicentre feasibility study that will investigate the use of a web application called SanaCoach Heart failure in patients with chronic heart failure. SanaCoach heart failure provides patient education, systematic self-monitoring, a care plan repository and facilitates correspondence with patient's care provider.

DETAILED DESCRIPTION:
Patients with chronic heart failure are encouraged to self-manage their illness, such as adhering to medical regimens, monitoring symptoms and adhere to lifestyle recommendations from the health care provider to optimise health outcomes and quality of life.

Consented study participants meeting the eligibility criteria for the STABILISE HF study will be using the the "SanaCoach heart failure" during a 6-month study period. SanaCoach heart failure is an application on the internet that supports patients and care providers in the development, implementation and monitoring of patient self-management. The SanaCoach heart failure provides information about heart failure, treatment, and lifestyle modifications. It can also monitor the patient's wellbeing, symptoms, vital signs, and gives advice on whether review with a health care provider is advisable. Furthermore, it provides a repository for patient's care plan to give insight into the course and treatment of the disorder.

Recruitment and dropout statistics will be assessed and the sociodemographic and comorbidity profile of consenting study participants as well as consenting non-participants (Patients who decide not to participate will be given an option to complete an anonymous sociodemographic survey.) will be analysed.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria in order to be eligible for this study.

* Adults (≥18 years) that own a device where SanaCoach heart failure can be used on
* Diagnosis of chronic heart failure according to ESC 2016 guidelines (HFrEF = LVEF <40%, HFmrEF = LVEF 40-49%, HFpEF = LVEF ≥ 50%), based on echocardiographic or MRI findings within the last year or considered stable before.
* Ability and willingness to give written informed consent and to comply with the requirements of the study

Exclusion Criteria:

Patients meeting any of the following criteria are NOT eligible for this study

* Patients without access to a device where SanaCoach heart failure can be used on
* Uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with participation in the clinical study, and/or put the subject at significant risk (according to investigator's [or delegate] judgment) if he/she participates in the clinical study.
* Patients that have been hospitalised for heart failure within the last 30 days.
* An underlying known disease, or surgical, physical, or medical condition that, in the opinion of the investigator (or delegate) might interfere with interpretation of the clinical study results.
* Treatment with other investigational products or devices within 30 days or five half-lives of the screening visit, whichever is longer.
* Planned use of other investigational products or devices during the course of the study.
* Any condition that according to the investigator could interfere with the conduct of the study, such as but not limited to:
* a. Subjects who are unable to communicate or to cooperate with the investigator.
* b. Unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
* c. Unlikely to comply with the protocol requirements, instructions, and study-related restrictions (eg, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study).
* d. Have any medical or surgical condition, which in the opinion of the investigator would put the subject at increased risk from participating in the study
* e. Persons directly involved in the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory heart failure patients evaluated in 4 different European sites
Sampling Method: Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Usability of the SanaCoach heart failure | Baseline to 6 months
  • Score on the System Usability Scale (SUS)

SECONDARY OUTCOMES:
Usability | Baseline to 6 months
  * % of users who rate SanaCoach heart failure as "easy to use"
  * % of users who rate SanaCoach heart failure as "transmits information as intended"
  * % of users who report satisfaction with the content of information received via SanaCoach heart failure
  * % of users motivated/intending to use SanaCoach heart failure
  * % of alerts/messages transmitted via the app that are rated "appropriate" by patient
  * % of alerts/messages transmitted via the app that are responded to appropriately by patient
Feasibility of the SanaCoach heart failure | Baseline to 6 months
  * Total number of hours of initial training on the use of SanaCoach heart failure attended by staff, patients, cardiologist
  * Total number of hours of refresher training on the use of SanaCoach heart failure attended by staff, patients, cardiologists
  * Total number of minutes/hours for patient counselling over study duration
  * Total number of minutes/hours spent on health record-keeping over study duration
Acceptability | Baseline to 6 months
  • Rate of completion of the intervention (i.e. number of participants who access and complete all aspects of the intervention including lifestyle coach support
Adherence rates | Baseline to 6 months
  • Number of completed/uncompleted education and monitoring sessions
Technology readiness index (TRI) | Baseline to 6 months
  Technology readiness index (TRI)

OTHER OUTCOMES:
Effectiveness | Baseline to 6 months
  * Number of unscheduled visits due to HF during the study period.
  * Number of cardiac rehospitalisation during the study period
Medication adherence | Baseline to 6 months
  • Changes in self-reported Medication adherence using the Medication Adherence Report Scale (MARS) from baseline to week 26.
Quality of life assessment | Baseline to 6 months
  • Changes in the Quality of life assessment with Kansas City Cardiomyopathy Questionnaire (KCCQ-12) from baseline to weeks 12 and 26.
Well-Being Index | Baseline to 6 months
  • World Health Organisation- Five Well-Being Index (WHO-5) from baseline to weeks 12 and 26.
Self-care Behaviour | Baseline to 6 months
  • Changes on the 9-Item European Heart Failure Self-care Behaviour Scale (EHFScB-9) from baseline to week 26.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Brunner-La Rocca, Prof, Principal Investigator — Maastricht University Medical Center
Locations (5):
- University Hospital Aachen, Aachen, Germany
- St. Michael's Hospital Dublin, Dublin, Ireland
- Maastricht UMC+, Maastricht, Netherlands
- United Kingdom (2):
  - Royal Victoria Hospital Belfast, Belfast
  - University of Suffolk, Ipswich

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon receipt of substantiated request to coordinator of the consortium.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the study. Expected Q2 of 2022
Access Criteria: Substantiated request to coordinator of the consortium with details about reason for request , which data and how the data will be used.

REFERENCES:
- [Derived] Gingele AJ, Amin H, De Wit K, Jacobsen M, Hageman A, van der Mierden K, Brandts J, Weerts J, Barrett M, Dixon LJ, Hill L, Knackstedt C, Brunner-La Rocca HP. Developing an artificial intelligence-based decision engine for disease-modifying therapy in heart failure: a pilot study. Eur Heart J Digit Health. 2023 Dec 1;6(2):285-288. doi: 10.1093/ehjdh/ztad075. eCollection 2025 Mar. PMID 40110213